CLINICAL TRIAL: NCT05171348
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of Multiple Ascending Doses of CM326 Injection by Subcutaneous Administration in Healthy Subjects
Brief Title: A Multiple Ascending Doses Study of CM326 Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM326HV002
Record Dates: First submitted 2021-12-09; First posted 2021-12-28 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2021-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CM326 55mg Q2W (Experimental): 55mg for 6 doses, SC, Q2W
  Interventions: Drug: CM326
- CM326 110mg Q2W (Experimental): 110mg for 6 doses, SC, Q2W
  Interventions: Drug: CM326
- CM326 220mg Q2W (Experimental): 220mg for 6 doses, SC, Q2W
  Interventions: Drug: CM326
- CM326 220mg Q4W (Experimental): 220mg for 3 doses, SC, Q4W
  Interventions: Drug: CM326
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CM326 — a humanized monoclonal antibody
  Arms: CM326 110mg Q2W; CM326 220mg Q2W; CM326 220mg Q4W; CM326 55mg Q2W
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, dose-escalating study to evaluate the safety, tolerability, PK profile, and immunogenicity of multiple SC administraion of CM326 at different doses in healthy subjects.

40 healthy male subjects will be enrolled in the study. The drug will be administered by dose-escalating principle at 4 dose levels: 55 mg Q2W, 110 mg Q2W, 220 mg Q2W, 220 mg Q4W.

ELIGIBILITY:
Inclusion Criteria:

* Male healthy volunteers, aged between 18 and 65 years of age inclusive, with a body mass index (BMI) within 18-26 kg/m2 (inclusive);
* Medical history, vital signs, physical examination, 12-lead Electrocardiogram, chest X-ray and abdominal color ultrasound are normal or abnormal with no clinical significance;
* All variables of clinical laboratory tests are normal or abnormal with no clinical significance;
* Subjects and partners agree to take effective contraception throughout the study (from screening to 3 months after the end of treatment);
* Capable of understanding the nature of the study and voluntarily signing the Informed Consent Form.

Exclusion Criteria:

* Known allergy to monoclonal antibody drugs or other related drugs, or allergy to excipients of CM326 injection;
* History of any clinically serious disease or history of circulatory, endocrine, neurological or hematological, immune, psychiatric, and metabolic diseases;
* History of asthma and allergic reactions;
* Use of any prescription drugs within 2 weeks prior to dosing, use of traditional Chinese medicine or over-the-counter drugs within 1 week prior to dosing;
* Received any marketed or investigational biologics within 5 half-lives (if known) or 12 weeks (whichever is longer) prior to dosing, or any investigational non-biologics within 5 half-lives (if known) or 4 weeks (whichever is longer) prior to dosing.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | up to Week 24
  Incidence of AEs, including any abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing.

SECONDARY OUTCOMES:
PK parameters: time to maximum concentration (Tmax). | up to Week 16
  Time to maximum concentration (Tmax).
PK parameters: maximum concentration (Cmax). | up to Week 16
  Maximum concentration (Cmax).
PK parameters: area under the plasma concentration-time curve over a dosing interval (AUCtau). | up to Week 16
  Area under the plasma concentration-time curve over a dosing interval (AUCtau).
PK parameters: area under the plasma concentration-time curve from 0 to t (AUC0-t). | up to Week 16
  Area under the plasma concentration-time curve from 0 to t (AUC0-t).
Immunogenicity endpoints: Occurrence of anti-drug antibodies (ADA) to CM326. | up to Week 16
  Occurrence of anti-drug antibodies (ADA) to CM326.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Di Y, Yang L, Zhou J, Zhang L, Huang Y, Jia Y, Yan H, Chen L, Hou Q, Chen B, Luo Z, Hou J. Translational Investigation of CM326 from Preclinical Studies to Randomized Phase I Clinical Trials in Healthy Adults. BioDrugs. 2025 May;39(3):487-498. doi: 10.1007/s40259-025-00714-4. Epub 2025 Apr 4. PMID 40185989